CLINICAL TRIAL: NCT05932810
Title: Evaluation of a Proactive Identification and Digital Mental Health Intervention Approach to Address Unmet Psychosocial Needs of Individuals Living With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Jennifer Dahne, Associate Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00126828
Record Dates: First submitted 2023-06-16; First posted 2023-07-06 (Actual); Results first posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Depression; Depressive Symptoms; Cancer
MeSH Terms: conditions — Depression; Neoplasms | interventions — Therapeutics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual (Other): Participants in the treatment as usual group will be provided educational material about mood management available via the EHR with the suggestion to discuss questions with their oncology provider. Participants will be asked to complete questionnaire measures weekly for 4 weeks following study enrollment.
  Interventions: Behavioral: Treatment as Usual
- Moodivate (Experimental): Participants randomized to the Moodivate condition will be instructed to utilize Moodivate regularly, at least once per day, for the treatment of depressed mood among cancer survivors. Participants in the Moodivate group will receive a download code to download the Moodivate mobile application. Moodivate is a mobile app for individuals with elevated symptoms of depression. Within the app, users identify values, create activities, schedule activities, and rate mood daily. Participants will be asked to complete questionnaire measures weekly for 4 weeks following study enrollment.
  Interventions: Behavioral: Behavioral Activation Therapy app

INTERVENTIONS:
Behavioral: Behavioral Activation Therapy app — Moodivate focuses on tracking daily activities, recording daily mood, and identifying new activities to complete that may help improve mood. Participants will be asked to complete questionnaire measures weekly for 8 weeks, with a final follow-up questionnaire at 12 weeks following study enrollment.
  Arms: Moodivate
Behavioral: Treatment as Usual — Participants will be provided educational material about mood management available via the EHR with the suggestion to discuss questions with their oncology provider. Participants will be asked to complete questionnaire measures weekly for 4 weeks following study enrollment.
  Arms: Treatment as Usual

SUMMARY:
The purpose of this research study is to evaluate a mobile application (app) for depression treatment called "Moodivate" among cancer survivors. Moodivate was developed by the investigators to assist with the treatment of depressed mood.

Participants will be randomly assigned to either download the mobile app, "Moodivate", or not. Approximately 2/3 of participants enrolled will receive the mobile app and the remaining 1/3 will not.

All participants will complete electronic questionnaire measures throughout the study period. Questionnaires will assess symptoms of depression, as well as the participant's experiences using Moodivate and participating in this trial. Participation in this study will take about 4 weeks, beginning today.

Participation in this study may help in the treatment of future cancer survivors. The greatest risks of this study include frustration, worsening of emotional distress, data breach, and/or loss of confidentiality. Alternative treatments include the participant contacting their primary care provider or their oncology care team to discuss other available treatments for depressed mood.

ELIGIBILITY:
Inclusion Criteria:

1. elevated depressive symptoms, defined as a score of ≥ 10 on the PHQ-936
2. ILLIC (as determined during manual chart review)
3. age 18+
4. currently own an iOS- or Android-compatible smartphone
5. report willingness to utilize a mobile app for the treatment of depressed mood (response of "yes" on yes/no item)
6. have a valid e-mail address that is checked regularly or have regular access to text messages (to access follow-up assessments)
7. English fluency

Exclusion Criteria:

1. Severe cognitive impairment that precludes completion of informed consent
2. current suicidal ideation on the PHQ-9 at screening or final study eligibility, defined as a response ≥1 (several days) on item nine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-05-05 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2024-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Dahne, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Graboyes EM, Levins O, DeMass R, Baskar N, Natale N, Sterba KR, Obeid JS, Sharma S, Hill EG, Dahne J. Proactive Identification and Digital Mental Health Intervention for the Treatment of Depression Among Individuals With Likely Incurable Cancer: A Pilot Randomized Clinical Trial. Psychooncology. 2025 Oct;34(10):e70309. doi: 10.1002/pon.70309. PMID 41125447

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment as Usual | Moodivate
Started | 10 | 20
Completed | 10 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment as Usual | Moodivate | Total
Number analyzed (Participants) | 10 | 20 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 14 | 22
  >=65 years | 2 | 6 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 2 | 10 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 20 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 8 | 15 | 23
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Accrual
Description: The proportion of Illic eligible for the trial who accrue to the study.
Time Frame: Study duration (6-7 months or until recruitment is reached)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment as Usual | Moodivate
Number analyzed (Participants) | 10 | 20
Participants | 10 | 20

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Treatment as Usual | Moodivate
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/20
Other Adverse Events (participants affected / at risk) | 0/10 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-04): https://cdn.clinicaltrials.gov/large-docs/10/NCT05932810/Prot_SAP_000.pdf